CLINICAL TRIAL: NCT05813366
Title: Combined Effect of Tryptophan Rich Diet and Acupuncture on Depression Related to Premenstrual Dysphoric Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Mohamed Ashour Gebril, Demonstrator at Physical Therapy department of Women's Health , Faculty of Physical Therapy, Horus University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003877
Record Dates: First submitted 2023-03-30; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Premenstrual Dysphoric Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tryptophan rich diet + vitamin B6 supplementation (Experimental): It will include 13 participants suffering from premenstrual dysphoric disorder (PMDD) who will be treated by diet rich wit tryptophan (high protein diet) for 8 weeks in addition to vitamin B6 tablets 60 mg once/day, throughout two menstrual cycles, starting from the first day of their menstrual cycle
  Interventions: Other: Tryptophan-Rich Diet; Other: Vitamin B6 Supplementation
- Acupuncture + Vitamin B6 supplementation (Experimental): It will include 13 participants suffering from premenstrual dysphoric disorder (PMDD) who will be treated by acupuncture twice a week for 8 weeks, resulting in a total of 16 visits. Each visit, including initial care, needle application and needle retention, will last about 45 min. In addition to vitamin B6 tablet 60mg once/day, throughout two menstrual cycles, starts from the first day of their menstrual cycle
  Interventions: Other: Acupuncture; Other: Vitamin B6 Supplementation
- Acupuncture + Tryptophan rich diet + vitamin B6 supplementation (Experimental): It will include 13 participants suffering from premenstrual dysphoric disorder (PMDD) who will be treated by diet rich with tryptophan (high protein diet) for 8 weeks and acupuncture twice a week for 8 weeks, resulting in a total of 16 visits. Each visit, including initial care, needle application and needle retention, will last about 45 min. In addition to vitamin B6 tablet 60mg once/day, throughout two menstrual cycles, starts from the first day of their menstrual cycle
  Interventions: Other: Acupuncture; Other: Tryptophan-Rich Diet; Other: Vitamin B6 Supplementation

INTERVENTIONS:
Other: Acupuncture — Tony disposable, single-use 0.20×40 mm Chinese needles will be used. The needle penetrates the skin sufficiently to reach the required depth and elicit de qi. The needles remains for 30 min, with gentle rotational movements applied three times during the session.
  Arms: Acupuncture + Tryptophan rich diet + vitamin B6 supplementation; Acupuncture + Vitamin B6 supplementation
Other: Tryptophan-Rich Diet — All participants in both groups (A and C) will be treated by high protein foods rich with tryptophan including: chicken , turkey, red meat, salmon, fish, tuna, beans, milk, cheese, seeds, nuts, egg, banana, kiwi, leafy greens, mushroom, broccoli and peas, etc.
  Total daily calorie intake will be calculated for each participant in both groups (A and C) before diet description. All females will serve the meals that met their required kilocalorie levels and physical activity levels so that the participants will not lose weight, feel hungry or be over-fed.
  Arms: Acupuncture + Tryptophan rich diet + vitamin B6 supplementation; Tryptophan rich diet + vitamin B6 supplementation
Other: Vitamin B6 Supplementation — All participants in all groups (A, B and C) will receive a tablet of vitamin B6 60mg once/day for 8 weeks, starting from the first day of their menstrual cycle, throughout two menstrual cycles.

SUMMARY:
Premenstrual Dysphoric Disorder (PMDD) is a severe form of premenstrual syndrome (PMS) affecting up to 8% of reproductive age women. It is characterized by physical and psychological symptoms that occur in the luteal phase of the menstrual cycle, prior to the onset of menses, and leads to negative impact on the psychosocial functioning of affected individuals.

Selective serotonin reuptake inhibitors are usually used to treat PMDD but they have several side effects so it is important to use complementary treatment such as tryptophan-rich diet and acupuncture for women with PMDD . The purpose of the current study is to determine the combined effect of tryptophan-rich diet and acupuncture on depression related to premenstrual dysphoric disorder

DETAILED DESCRIPTION:
This study will be conducted on 39 participants suffering from premenstrual dysphoric disorder (PMDD). They will be recruited from Horus University, New Damietta, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* All females will be clinically diagnosed with premenstrual dysphoric disorder (PMDD) as confirmed and referred from the gynaecologist.
* All females will be firstly assessed by Hamilton Depression rating scale (HDRS) for two months to confirm depression related to PMDD before participating in the study.
* Their ages will be ranged from 20 to 30 years.
* Their BMI will be ranged from 20 to 25 kg/m.
* Being virgin.
* Having regular menstruation for the last 6 months (every 28- 35 days with no intermittent bleeding).
* All females have a sedentary lifestyle.
* Voluntary acceptance of participation in the study

Exclusion Criteria:

* Using hormonal contraception (such as oral contraceptives and injections).
* Menstrual irregularity.
* Using diuretics or psychiatric medications.
* Using chronic non-steroidal anti-inflammatory drugs.
* Pre-diagnosed with any other psychological problems not related to PMDD.
* Follow any exercise programs.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-04-25 (Estimated); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
The Premenstrual Symptoms Screening Tool (PSST) | Up to 2 months
  It is a validated, simple, user-friendly screening tool to identify women who suffer from severe Premenstrual Syndrome (PMS) or Premenstrual Dysphoric Disorder (PMDD). It reflects and 'translates' categorical Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria into a rating scale with degrees of severity (Not at all, mild, moderate, severe). The scoring will be as follows:
  the following criteria must be present for a diagnosis of PMDD:
  * At least one of #1, #2, #3, and #4 is severe.
  * In addition at least four of #1 - #14 are moderate to severe.
  * At least one of A, B, C, D and E is severe.
Hamilton Depression Rating Scale (HDRS) | Up to 2 months
  The HDRS (also known as the Ham-D) is the most widely used clinician-administered depression assessment scale. HRSD provides a reliable and valid assessment of depression.
  Method for scoring varies by version. For the HDRS17, a score of 0 - 9 is generally accepted to be within the normal range, 10 - 13 mild, 14-17 mild to moderate and >17 moderate to severe

SECONDARY OUTCOMES:
Quality of Life Enjoyment and Satisfaction Questionnaire - short form | Up to months 2
  It evaluates overall enjoyment and satisfaction with physical health, mood, work, household and leisure activities, social and family relationships, daily functioning, sexual life, economic status, overall well-being and medications.
  Responses are scored on a 5-point scale ("very poor" to "very good"), where higher scores indicate better enjoyment and satisfaction with life (possible range 14-70). Previous study had shown that it is reliable, valid and sensitive assessments of the individuals' quality of life (QOL)